CLINICAL TRIAL: NCT04246346
Title: Effectiveness of Using Interactive Consulting System Based on Large Language Model to Enhance Informed Choice of Cataract Patients: a Non-inferiority Randomized Controlled Trial
Brief Title: Effectiveness of Using Interactive Consulting System to Enhance Informed Choice
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yingfeng Zheng, Clinical Investigator, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 2020KYPJ003
Record Dates: First submitted 2020-01-23; First posted 2020-01-29 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Age-related Cataract

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interactive chatbot (Experimental): A chatbot embedded into a mobile application which is able to bidirectionally interact with patients and provide standard general information, quantitative risk information on the possible outcomes of cataract surgery.
  Interventions: Other: An interactive chatbot for patient decision aid
- Senior ophthalmologists (Active Comparator): Senior ophthalmologists would communicate with patients and provide standard general information, quantitative risk information on the possible outcomes of cataract surgery.
  Interventions: Other: Senior ophthalmologists

INTERVENTIONS:
Other: An interactive chatbot for patient decision aid — A chatbot embedded into a mobile application which is able to bidirectionally interact with patients and provide standard general information, quantitative risk information on the possible outcomes of cataract surgery.
  Arms: Interactive chatbot
Other: Senior ophthalmologists — Senior ophthalmologists would communicate with patients and provide standard general information, quantitative risk information on the possible outcomes of cataract surgery.
  Arms: Senior ophthalmologists

SUMMARY:
To compare the performance of an interactive chatbot versus senior ophthalmologists for enhancing informed decisions made by cataract patients. The chatbot was built based on large language models, and could generate medical expert-level responses.

DETAILED DESCRIPTION:
Cataract surgery is the only way to treat age-related cataract. For patients at early or moderate stages, cataract surgery is an elective surgery without objective indications. Therefore the patients are uaually not aware whether they should receive the surgery. The number of trained and qualified ophthalmologists are limited in China and lots of patients cannot have detailed consultation with ophthalmologists. As a result, many patients still have doubts about whether they should receive cataract surgery or not. In this study, we aim to assess the effectiveness of an interactive chatbot based on large language models versus senior ophthalmologists to enhance informed decisions made by cataract patients.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals aged 45-80 years who have been resident in the selected study district for more than six months;
2. A definite diagnosis of age-related cataract;
3. Having not received cataract surgery;
4. Willing to participate the study and provide informed consent.

Exclusion Criteria:

1. Bilateral blindness (presenting distance visual acuity worse than 3/60);
2. Having ocular, hearing or mental disorders precluding reading or telephone interview;
3. Ocular disorders other than cataract leading to permanent vision loss that could not be corrected through cataract surgery;
4. Having cataract surgery contraindication.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 660 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Informed choice about cataract surgery (the proportion of participants who make an informed choice，which is defined as a good knowledge score and an intention that is consistent with their attitude score) | 2 weeks post intervention
  Informed choice is an aggregated measure of multiple measurements, including knowledge (a 12-item questionnaire that assesses conceptual (items 1-10) and numerical (items 11-12) knowledge), attitudes (6 items, with 5 responses for each), and intentions (single item with 5 responses)

CONTACTS AND LOCATIONS:
Overall Officials: Yingfeng Zheng, MD, PhD, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhognshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Deidentified will be shared after the study being published.
Supporting Information: Study Protocol, ICF
Time Frame: The data will be available upon request after the study being accepted by peer-reviewed journal and published online.
Access Criteria: The data will be available upon request. Requestors will be asked to sign data sharing agreements.